CLINICAL TRIAL: NCT02559089
Title: Multicenter and Prospective Clinical Registry Study of Anti-N-methyl-D-aspartate Receptor Encephalitis in China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Xuanwu Hospital, Beijing (Other); Peking Union Medical College Hospital (Other); Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Jia Wei Wang,MD, Chairman and Full Professor of Department of Neurology and Medical Research Center, Beijing Tongren Hospital
Other Study IDs: 2014-1-1101-1
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Anti-NMDA Receptor Enphalitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- anti-NMDA receptor encephalitis
- other autoimmune encephlitis
- other encephalopathy

SUMMARY:
Anti-NMDA receptor encephalitis is the most common curable non-infectious autoimmune encephalitis，but because of the lack of recognition in the clinic, usually been misdiagnosed as other causes of encephalitis. Therefore, it is urgent to establish a database of anti-NMDA receptor encephalitis in Chinese population. The multi-center, prospective clinical trial of anti-NMDA receptor encephalitis in China's , combined with Beijing Xuanwu hospital, Beijing Tiantan Hospital, Beijing Children's Hospital and other hospitals around the country, by screening the NMDA receptor antibody and summarizing the cases analysis, in order to provide evidence for clinical diagnosis and treatment of anti-NMDA receptor encephalitis.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 6 months.
2. Encephalopathy symptoms (change of mental state and consciousness level) persist for more than 24 hours;
3. At least one or more clinical features of the followings: fever, epilepsy, focal neurological deficiency symptoms, changes in CSF(cerebrospinal fluid inflammatory), changes in EEG (electroencephalogram), radiographic abnormalities;
4. Clinical suspected encephalitis, but conventional detected methods cannot make etiology clear.
5. Signed informed consent

Exclusion Criteria:

1. Infants less than 6 months;
2. The metabolic encephalopathy;
3. Infectious encephalitis with clear pathogen clinically, referring the specific pathogenic microorganisms, including: bacteria, virus, fungus, parasite, spirochete and so on;
4. Non-infectious encephalitis with clear diagnosis clinically, including: multiple sclerosis, neuromyelitis optic, acute disseminated encephalomyelitis and so on.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the unidentified encephalitis patients who meeting the inclusion criteria and exclusion criteria and signing the written informed consent form。
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
death | 30 days